CLINICAL TRIAL: NCT04996082
Title: Skin Fibrosis Analysis by Raman Spectroscopy in Systemic Sclerosis
Acronym: RAMSES
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO21044
Record Dates: First submitted 2021-08-03; First posted 2021-08-09 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Validation of Raman Spectroscopy Usefulness in Systemic Sclerosis
Keywords: Systemic sclerosis; Raman spectroscopy
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Systemic sclerosis group: Patients with systemic sclerosis
- No Systemic sclerosis group: Patients without systemic sclerosis

SUMMARY:
Systemic sclerosis (SSc) is a rare connective tissue disease characterized by a high clinical heterogeneity with unpredictable evolution that could engage functional and life-threatening prognosis. Most of patients develop skin fibrosis gradually spreading. Two clinical distinct forms are described according to the extension of skin fibrosis: limited (lSSc) and diffuse (dSSc) SSc. It is now admitted that a spreading of skin fibrosis is associated with poor prognosis. This disease can be complicated by pulmonary arterial hypertension (PAH), interstitial lung disease (ILD) and scleroderma renal crisis (SRC) representing the main causes of death in SSc. Usually, PAH is associated with lSSc, and ILD and SRC are associated with dSSc. Prognosis is also different regarding skin phenotype with a higher mortality rate in dSSc.

An easy score, called modified Rodnan skin score, is commonly used in clinical practice to evaluate the spreading and severity of skin fibrosis, but this score is hardly reproducible. Ultrasound can be used to measure skin thickness and is more reproducible than the Rodnan skin score. Nevertheless, non-invasive analysis of fibrosis composition in different areas is not possible with these two technics.

Thus, in this study we will investigate Raman spectroscopy, a non-invasive technic based on the interaction of a low-intensity laser with matter.

DETAILED DESCRIPTION:
Raman spectroscopy will be performed on patients with SSc, according to the ACR criteria, and control patients without SSc, on 3 different areas of the skin. Patients with SSc and controls will be matched by gender and age. These measures will be performed at 6 months, 12 months, 24 months and 36 months.

ELIGIBILITY:
inclusion criteria :

* patients with SSc, according to ACR criteria
* older than 18-years-old exclusion criteria :
* younger than 18-years-old
* patient protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with or without systemic sclerosis, according to ACR criteria, older than 18-years-old
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Raman spectroscopy | at 6 months
Raman spectroscopy | at 12 months
Raman spectroscopy | at 24 months
Raman spectroscopy | at 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France